CLINICAL TRIAL: NCT02871102
Title: Right-Sizing Tidal Volume in ARDS: Using the Stress Index to Optimize Mechanical Ventilation to Individual Respiratory Mechanics
Brief Title: Stress Index to Individualize Mechanical Ventilation in ARDS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The ART Trial was published suggesting harm by the intervention protocol, which was closely related to the protocol in this study, so the study was terminated.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Andrew McKown, Fellow in Pulmonary and Critical Care Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 160770
Record Dates: First submitted 2016-08-10; First posted 2016-08-18 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: mechanical ventilation; respiratory mechanics; acute respiratory distress syndrome; positive end-expiratory pressure; tidal volume
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Arm (Experimental)
  Interventions: Procedure: Recruitment Maneuver with PEEP and Tidal Volume Optimization

INTERVENTIONS:
Procedure: Recruitment Maneuver with PEEP and Tidal Volume Optimization — A staircase recruitment maneuver will be performed on pressure control ventilation followed by a decremental PEEP trial. During the decremental PEEP trial inspiratory tidal volumes will be varied at each step between 3 ml/kg and 10 ml/kg predicted body weight while recording the continuous pressure and flow tracings from the mechanical ventilator. With each PEEP and tidal volume combination, end expiratory and end-inspiratory plateau pressure and stress index will be assessed. At the completion of the decremental PEEP trial, the patient will be returned to ARDSnet-recommended ventilator settings.

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a widely prevalent and morbid disease for which the current standard treatment is supportive care and avoidance of complications with lung-protective ventilation. Lower-tidal volume ventilation has been largely accepted as a means of lung protective ventilation, but the mechanism for its effectiveness is not yet clear, and debate remains as to how best to choose positive end-expiratory pressure (PEEP). Reduction in driving pressure (plateau pressure minus PEEP) has been suggested as a possible means to minimize ventilator-induced lung injury. This protocol aims to identify the range of safe paired-settings of PEEP and tidal volume, with selection guided by driving pressure and the stress index, a tool to recognize potential lung hyperinflation during mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Intensive Care Unit
* Receiving invasive mechanical ventilation via endotracheal or tracheostomy tube
* Presence of ARDS by Berlin Criteria (acute onset bilateral pulmonary infiltrates incompletely explained by left heart failure together with a PaO2/FiO2 of <300 or SpO2/FiO2 <315)

Exclusion Criteria:

* Inability to obtain surrogate consent
* Presence of specified comorbidities:

  1. pregnancy
  2. pre-existing severe chronic obstructive pulmonary disease, defined as FEV1 documented < 1L or baseline hypercapnia
  3. cerebral edema
  4. known intra-cranial abnormality
  5. acute coronary syndrome
* Endotracheal or tracheostomy cuff leak
* Chest tube with persistent air leak
* Severe hemodynamic instability (defined as attending judgment that the patient is unable to safely tolerate ventilator manipulations)
* Presence of spontaneous respiratory activity as evidenced by examination of the ventilator waveform tracing
* Intrinsic PEEP of > 5 cmH2O
* Assessment of study staff or patient's attending physician that the patient would not be a good study participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Comparison of ARDSnet-optimized and protocol-optimized tidal volume | Completion of the study intervention, less than 1 day
  Mean absolute difference between tidal volume in cc/kg PBW prescribed by ARDSnet settings on ARDSnet PEEP versus maximal protective tidal volume defined by stress index <1.05 at the ARDSnet PEEP on experimental protocol.
Comparison of ARDSnet-optimized and protocol-optimized driving pressure | Completion of the study intervention, less than 1 day
  Mean difference in driving pressure prescribed by ARDSnet settings versus at lowest measured possible driving pressure that achieves equivalent minute ventilation as ARDSnet table with respiratory rate < or = 35 per minute and SI <1.05.

SECONDARY OUTCOMES:
Comparison of ARDSnet-optimized and protocol-optimized PEEP | Completion of the study intervention, less than 1 day
  Mean absolute difference between safest PEEP as determined by experimental protocol with tidal volume of 6 mL/kg PBW (defined as the PEEP at which 6 mL/kg PBW yields the lowest driving pressure with a SI <1.05) versus the PEEP established by ARDSnet table.
Comparison of ARDSnet-optimized and protocol-optimized elastance | Completion of the study intervention, less than 1 day
  Mean difference in elastance prescribed by ARDSnet settings versus at lowest measured possible elastance achieving equivalent minute ventilation as ARDSnet table with respiratory rate < or = 35 per minute.

OTHER OUTCOMES:
ICU-free days to 14 days after enrollment | 14 days post-enrollment
  Comparison of ICU-free days to 14 days after enrollment between groups of those patients who are ventilated with settings that coincide with those determined to be most protective by the experimental protocol (within 0.5 cc/kg PBW tidal volume and 1 cmH2O of PEEP) versus those not.
Ventilator-free days to 14 days after enrollment | 14 days post-enrollment
  Comparison of ventilator-free days to 14 days after enrollment between groups of those patients who are ventilated with settings that coincide with those determined to be most protective by the experimental protocol (within 0.5 cc/kg PBW tidal volume and 1 cmH2O of PEEP) versus those not.
ICU mortality at 28 days | 28 days post-enrollment
  Comparison of 28-day ICU mortality post-enrollment between groups of those patients who are ventilated with settings that coincide with those determined to be most protective by the experimental protocol (within 0.5 cc/kg PBW tidal volume and 1 cmH2O of PEEP) versus those not.
In-hospital mortality at 28 days | 28 days post-enrollment
  Comparison of 28-day in-hospital mortality post-enrollment between groups of those patients who are ventilated with settings that coincide with those determined to be most protective by the experimental protocol (within 0.5 cc/kg PBW tidal volume and 1 cmH2O of PEEP) versus those not.
Time-varying elastance | Completion of the study intervention, less than 1 day
  Assessment of the stability of a model-imputed estimate of time-varying elastance for a given insufflation volume independent of total tidal volume per breath.
Comparison of ARDSnet-optimized and time-varying elastance-optimized tidal volume | Completion of the study intervention, less than 1 day
  Mean absolute difference between tidal volume in cc/kg PBW prescribed by ARDSnet settings on ARDSnet PEEP versus maximal protective tidal volume defined by the point of rise of model-imputed time-varying elastance at ARDSnet PEEP on experimental protocol.
Comparison of ARDSnet-optimized and time-varying elastance-optimized driving pressure | Completion of the study intervention, less than 1 day
  Mean difference in driving pressure prescribed by ARDSnet settings versus at lowest measured possible driving pressure that achieves equivalent minute ventilation as ARDSnet table with respiratory rate < or = 35 per minute and time-varying elastance not rising.
Comparison of ARDSnet-optimized and time-varying elastance-optimized PEEP | Completion of the study intervention, less than 1 day
  Mean absolute difference between safest PEEP as determined by experimental protocol with tidal volume of 6 mL/kg PBW (defined as the PEEP at which 6 mL/kg PBW yields the lowest driving pressure without a rising time-varying elastance) versus the PEEP established by ARDSnet table.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] McKown AC, Semler MW, Rice TW. Best PEEP trials are dependent on tidal volume. Crit Care. 2018 May 2;22(1):115. doi: 10.1186/s13054-018-2047-4. PMID 29720277